CLINICAL TRIAL: NCT07153003
Title: Efficacy And Safety Of Tramadol And Oxycodone Versus Oxycodone Monotherapy For Pain Control After Primary Total Knee And Total Hip Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: Efficacy And Safety Of Tramadol And Oxycodone Versus Oxycodone Monotherapy For Pain Control After Primary Total Knee And Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles P. Hannon, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-002295
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Oxycodone; Tramadol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxycodone Only (Active Comparator): Patient's will be prescribed only Oxycodone for post operative pain management.
  Interventions: Drug: Oxycodone
- Multimodal Pain Control (Active Comparator): Patients will be prescribed Tramadol and Oxycodone for post operative opioid pain relief.
  Interventions: Drug: Tramadol and Oxycodone

INTERVENTIONS:
Drug: Oxycodone — Patients will receive oral Oxycodone only to treat post-operative pain:
  Oxycodone 5mg
  * Patients ≤75 years old: 5mg or 10 mg PO every 4 hr as needed
    * 5 mg for pain rated 4-6
    * 10 mg for pain rated 7-10
  * Patients >75 years old and/or sensitive to opioids or sedatives: 2.5mg or 5mg every 4hr as needed
    * 2.5mg for pain rated 4-6
    * 5mg for pain rated 7-10
  Arms: Oxycodone Only
Drug: Tramadol and Oxycodone — Patients will receive a combination of Tramadol and Oxycodone to take orally to treat post-operative pain:
  Tramadol 50mg
  * Patients ≤75 years old: 50 mg for pain rated 4-6; 100 mg for pain rated 7-10
  * Patients >75 years old and/or sensitive to opioids or sedatives; use 50 mg
  * Dosing is every 8 hours as needed. Cumulative dose not to exceed 400mg in 24 hours
  Oxycodone 5mg
  * Patients ≤75 years old: 5mg or 10 mg PO every 4 hr as needed if still having pain after maximum tramadol administration
    * 5 mg for pain rated 4-6
    * 10 mg for pain rated 7-10
  * Patients >75 years old and/or sensitive to opioids or sedatives: 2.5mg or 5mg every 4 hr as needed if still having pain after maximum tramadol administration
    * 2.5 mg for pain rated 4-6
    * 5 mg for pain rated 7-10
  Arms: Multimodal Pain Control

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of tramadol and oxycodone therapy in comparison to oxycodone alone as part of a multimodal pain regimen to reduce postoperative opioid consumption, pain, minimize adverse events and complications for primary total knee arthroplasty (TKA) and primary total hip arthroplasty (THA).

ELIGIBILITY:
Inclusion Criteria:

* Primary TKA
* Primary THA
* Age > 18 years

Exclusion Criteria:

* Age < 18 years
* Revision or partial TKA/THA
* Pregnant or breast-feeding women
* Simultaneous bilateral TKA/THA
* Primary TKA/THA due to oncologic reason
* Anaphylaxis to opioids
* Renal or liver failure
* Prior opioid use disorder/ substance use disorder
* Opioid use within 3 months prior to surgery
* Patients needing a translator and those with dementia or other cognitive deficits
* Patients taking Monoamine Oxidase Inhibitor (MOAI) medications (phenelzine, tranylcypromine) or benzodiazepine medications (alprazolam, diazepam, lorazepam, etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2031-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption during the first 30 days | 30 days
  Total amount of opioid medication taken for the first 30 days following surgery, reported in milligrams (mg)

SECONDARY OUTCOMES:
Cumulative opioid consumption during the first 90 days | 90 days
  Total amount of opioid medication taken for the first 90 days following surgery, reported in milligrams (mg)
Postoperative opioid refills within 90 days | 90 days
  Total number of opioid medication refills within 90 days post surgery
Number of unused opioid pills | 90 days
  Total number of unused opioid pills unused after 90 days
Change in Visual Analogue Scale (VAS) pain scores | Daily for 90 days
  Pain values reported by participants will be assessed using the 100-mm Visual Analogue Scale (VAS). The VAS line will be 100 mm long with no intermediate delineations. Each end will be marked with "no pain" on the left, and "worst possible pain" on the right. Participants will identify their pain level by indicating a point on the line between each end. That point will be measured from the "No pain" end, and the number of millimeters will be reported as the pain score.
Number of complications | 90 days
  Total number of complications experienced post-operatively, complications include stiffness, VTE, GI hemorrhage, falls, ileus, dizziness, changes in vision, and miosis.
Number of emesis episodes | 90 days
  Postoperative nausea and vomiting will be measured by total number of emesis episodes
Rate of antiemetic use | 90 days
  Total number of times patients require use of antiemetics for nausea or vomiting
Satisfaction survey scores | 90 days
  Patients will be provided with a satisfaction survey 90 days post-surgery. The survey consists of 2 questions rated on a Likert scale measuring understanding and confidence in medication use, and one yes/no question. The Likert scale questions are ranked from "0" - no understanding/low confidence to "10" - full understanding/high confidence. Higher scores indicate greater satisfaction with the prescribed opioid therapy plan.
Length of Stay | Post-operatively, up to 90 days
  Total number of days patients stay inpatient

CONTACTS AND LOCATIONS:
Overall Officials: Charles P. Hannon, MD, MBA, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials